CLINICAL TRIAL: NCT00813527
Title: A Double-blind, Randomized Study to Evaluate the Efficacy and Safety of TAK-475 or Placebo When Coadministered With Fenofibrate in Subjects With Combined Hyperlipidemia
Brief Title: Effect of Lapaquistat Acetate Combined With Fenofibrate on Blood Cholesterol Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-05-TL-475-031; U1111-1122-8178 (Registry Identifier: WHO)
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Hyperlipidemias
Keywords: Drug Therapy; Lipid Metabolism Disorders; Hyperlipidemias; Hypercholesterolemia; Hypertriglyceridemia
MeSH Terms: conditions — Hyperlipidemias; Lipid Metabolism Disorders; Hypercholesterolemia; Hypertriglyceridemia | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lapaquistat Acetate 100 mg QD + Fenofibrate 145 mg QD (Experimental)
  Interventions: Drug: Lapaquistat acetate and fenofibrate
- Fenofibrate 145 mg QD (Active Comparator)
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: Lapaquistat acetate and fenofibrate — Lapaquistat acetate 100 mg, tablets, orally, once daily and fenofibrate 145 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: Lapaquistat; TAK-475
  Arms: Lapaquistat Acetate 100 mg QD + Fenofibrate 145 mg QD
Drug: Fenofibrate — Lapaquistat acetate placebo-matching tablets, orally, once daily and fenofibrate 145 mg, tablets, orally, once daily for up to 12 weeks.
  Other Names: Tricor; Trilipix
  Arms: Fenofibrate 145 mg QD

SUMMARY:
The purpose of this study is to compare changes in cholesterol levels in patients with elevated blood cholesterol with administration of lapaquistat acetate, once daily (QD), and fenofibrate.

DETAILED DESCRIPTION:
Elevated plasma cholesterol (hypercholesterolemia) and various other plasma lipid imbalances (dyslipidemias) are major risk factors for coronary heart disease. It has been established that lowering the low-density lipoprotein cholesterol plasma concentration effectively reduces cardiovascular morbidity and mortality. As a result of this finding, the National Cholesterol Education Program Adult Treatment Panel III identifies control of low-density lipoprotein cholesterol as essential in the prevention and management of coronary heart disease.

Currently, 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitors (statins) are the first-line monotherapies prescribed to reduce low-density lipoprotein cholesterol, after diet and therapeutic lifestyle change. However, low doses of statins often fail to produce the Adult Treatment Panel III-recommended levels of low-density lipoprotein cholesterol reduction, making it necessary to increase the dose or add an additional treatment. This in turn may result in decreased tolerability and potential safety concerns.

At higher doses, statins are associated with various myopathies ranging from rare occurrences of rhabdomyolysis and myositis to more frequent symptoms of muscle weakness, cramps, or pain; these can occur with mild or no increases in creatine kinase. Statin use also is associated with increases in liver transaminase levels. These tolerability and safety concerns may contribute to the high discontinuation rates of statins and their prescription at low, and often ineffective, doses.

TAK-475 (lapaquistat acetate) inhibits the cholesterol synthesis pathway at a different step than statins (acting on squalene synthase rather than 3-hydroxy-3-methylglutaryl coenzyme A); it does not reduce concentrations of isoprenylated intermediates believed to be responsible for the myopathies associated with statin use.

This study was conducted to determine whether lapaquistat acetate with fenofibrate has the potential to be more effective than fenofibrate by itself in lowering low-density lipoprotein cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing potential must not be pregnant as determined by a negative serum human chorionic gonadotropin, not lactating, not planning on becoming pregnant between Screening and 30 days following the last dose of study medication, and agreed to use acceptable forms of contraception during the study.
* Prior to Randomization, must have a mean low density lipoprotein cholesterol greater than or equal to 100 mg/dL (2.59 mmol/L) for 2 consecutive samples. The difference between the two individual low density lipoprotein cholesterol values not to exceed 15% of the higher value.
* Prior to Randomization, must have mean triglycerides greater than or equal to 150 and less than or equal to 600 mg/dL (1.70 and 6.78 mmol/L, respectively) for 2 consecutive samples. The upper value for either triglycerides sample must have been less than or equal to 650 mg/dL (7.35 mmol/L).
* Clinical laboratory evaluations (including clinical chemistry [fasted for at least 10 hours], hematology and urinalysis) within the reference range for the testing laboratory unless results deemed not clinically significant or considered within normal limits for this subject by the investigator or the sponsor.
* Willing and able to continue to comply with a standardized low cholesterol diet.

Exclusion Criteria:

* Alanine aminotransferase or aspartate aminotransferase level of greater than 1.5 times the upper limit of normal, active liver disease or jaundice.
* Serum creatinine greater than 1.5 mg/dL (133 μmol/L).
* Creatine phosphokinase greater than 3 times the upper limit of normal.
* Diabetes with a hemoglobin A1c greater than 8 % at Visit 1.
* Previous history of cancer in remission for less than 5 years prior to the first dose of study medication. Does not include those subjects with basal cell or stage I squamous cell carcinoma of the skin.
* An endocrine disorder, such as Cushing's syndrome, hyperthyroidism, or inappropriately treated hypothyroidism, affecting lipid metabolism. Subjects with hypothyroidism on appropriate replacement therapy (defined as stable thyroid hormone replacement therapy at least 3 months prior to Visit 1 and thyrotropin levels less than 1.5 times the upper limit of normal) are eligible for enrollment. If thyrotropin is greater than 1.5 times upper limit of normal, a free thyroxine level is to be determined. If the free thyroxine is within normal limits for that subject, the subject may continue in the study.
* History of myocardial infarction, unstable angina, transient ischemic attacks, cerebrovascular accident, percutaneous coronary intervention, coronary or peripheral arterial surgery (bypass graft surgery) in the 6 months prior to Visit 1.
* Positive hepatitis B surface antigen, or hepatitis C virus antibody, as determined by medical history and/or subject's verbal report.
* Positive human immunodeficiency virus status or is taking anti-retroviral medications, as determined by medical history and/or subject's verbal report.
* Unable or unwilling to discontinue excluded medications or to continue stable doses of "stable dose" medications or required treatment with any excluded medication during the study.
* Exposure to TAK-475 in other studies or currently is participating in another investigational study or has participated in an investigational study within the past 30 days or, for drugs with a long half-life, within a period of less than 5 times the drug's halflife.
* Known hypersensitivity or history of adverse reaction to any fibrate.
* History or presence of clinically significant food allergy that would prevent adherence to the therapeutic lifestyle change (or equivalent) diet.
* Known homozygous familial hypercholesterolemia or known Type III hyperlipoproteinemia (familial dysbetalipoproteinemia).
* Active cholecystitis or known cholelithiasis (a fibrate risk factor).
* Severe renal or hepatic dysfunction, including biliary cirrhosis during Run-In or at Randomization (a fibrate risk factor).
* Fibromyalgia, myopathy, rhabdomyolysis or unexplained muscle pain.
* Uncontrolled hypertension (defined as resting diastolic blood pressure greater than100 mm Hg or resting systolic blood pressure greater than 160 mm Hg) at Visit 1.
* Inflammatory bowel disease or any other malabsorption syndrome or has had gastric bypass or any other surgical procedure for weight loss.
* Unwilling or unable, in the opinion of the investigator, to comply with the protocol or scheduled appointments.
* Unable to understand verbal or written English or any other language for which a certified translation of the approved informed consent was available.
* History of drug abuse (defined as illicit drug use) or a history of alcohol abuse (defined as regular or daily consumption of more than 2 alcoholic drinks per day) within the past 2 years.
* Any other serious disease or condition at Screening or at Randomization that might reduce life expectancy, impair successful management according to the protocol, or make the subject an unsuitable candidate to receive study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2006-02; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Percent change from Baseline in direct fasting plasma low-density lipoprotein cholesterol. | Week 12 or Final Visit.

SECONDARY OUTCOMES:
Change from baseline in calculated low-density lipoprotein cholesterol. | Week 12 or Final Visit.
Change from baseline in non- high-density lipoprotein cholesterol. | Week 12 or Final Visit.
Change from baseline in total cholesterol. | Week 12 or Final Visit.
Change from baseline in apolipoprotein B. | Week 12 or Final Visit.
Change from baseline in triglycerides. | Week 12 or Final Visit.
Change from baseline in high-density lipoprotein cholesterol. | Week 12 or Final Visit.
Change from baseline in apolipoprotein A1. | Week 12 or Final Visit.
Change from baseline in very-low-density lipoprotein cholesterol. | Week 12 or Final Visit.
Change from baseline in derived ratios including total cholesterol/high-density lipoprotein cholesterol, low-density lipoprotein cholesterol/high-density lipoprotein cholesterol, and apolipoprotein B/ apolipoprotein Al. | Week 12 or Final Visit.
Change from baseline in high-sensitivity C-reactive protein. | Week 12 or Final Visit.
Percentage of Subjects Achieving Target Direct low-density lipoprotein cholesterol Levels. | Week 12 or Final Visit.

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Takeda
Locations (36):
- United States (32):
  - Huntsville, Alabama
  - Sierra Vista, Arizona
  - Beverly Hills, California
  - Long Beach, California
  - Spring Valley, California
  - Colorado Springs, Colorado
  - Golden, Colorado
  - Waterbury, Connecticut
  - Jacksonville, Florida
  - Kissimmee, Florida
  - Miami, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Pinellas Park, Florida
  - West Palm Beach, Florida
  - Warner Robins, Georgia
  - Chicago, Illinois
  - Peoria, Illinois
  - Indianapolis, Indiana
  - Wichita, Kansas
  - Edina, Minnesota
  - St Louis, Missouri
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Hillsboro, Oregon
  - Beaver, Pennsylvania
  - Goose Creek, South Carolina
  - Nashville, Tennessee
  - Norfolk, Virginia
  - Richmond, Virginia
- Canada (4):
  - Coquitlam, British Columbia
  - Victoria, British Columbia
  - London, Ontario
  - Toronto, Ontario

REFERENCES:
- [Result] Stein EA, Bays H, O'Brien D, Pedicano J, Piper E, Spezzi A. Lapaquistat acetate: development of a squalene synthase inhibitor for the treatment of hypercholesterolemia. Circulation. 2011 May 10;123(18):1974-85. doi: 10.1161/CIRCULATIONAHA.110.975284. Epub 2011 Apr 25. PMID 21518985